CLINICAL TRIAL: NCT00770198
Title: Study of IL-6 Transsignaling in Chronic Human Liver Disease
Brief Title: sgp130 in Chronic Human Liver Disease
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Olivier Le Moine, MD, PhD, Erasme University Hospital
Other Study IDs: AL-gp130
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2008-10-09 (Estimated); Status verified 2008-10

CONDITIONS: Alcoholic Liver Disease; Chronic Hepatitis C Virus Infection
Keywords: liver; alcohol; HCV
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma, liver biopsies, and peripheral blood mononuclear cell culture medium.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- alcoholic liver disease: alcoholic liver disease patients undergoing a transjugular liver biospy in our institution
- chronic HCV hepatitis: chronic HCV hepatitis patients undergoing a transjugular liver biopsy in our institution

SUMMARY:
Chronic liver disease are characterized by increased levels of plasma IL-6, but the bioactivity of this cytokine in this disease is not well known. IL-6 receptor complex is regulated by multiple receptors subunits: the soluble form of IL-6 Receptor enhance IL-6 signal by a process called trans-signaling on cells expressing few membrane IL-6 receptors. Soluble gp130 is the natural inhibitor of IL-6 trans-signaling. The aim of this study is to characterize circulating and liver levels of theses compounds of IL-6 receptor complex, to unravel the bioactivity of IL-6 in this disease.

DETAILED DESCRIPTION:
Consecutive patients undergoing transjugular liver biopsies for alcoholic liver disease or hepatitis C virus infection will be included in the study to measure plasma cytokines levels, peripheral blood mononuclear cells cytokine release and liver IL-6R compounds mRNA levels.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol excess intake and suspected liver disease
* Alcohol excess intake and clinical liver cirrhosis
* chronic hepatitis C virus infection and suspected liver disease
* chronic hepatitis C virus infection and clinical liver cirrhosis

Exclusion Criteria:

* other (superimposed) liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients of Erasme University Hospital
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2005-01; Primary Completion 2007-01 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Lemmers, MD, Principal Investigator — Erasme Hospital, Gastroenterology Dpt
Locations (1):
- Hopital Erasme - Dpt of Gastroenterology, Brussels, Belgium